CLINICAL TRIAL: NCT03277365
Title: MyGeneRank: A Digital Platform for Next-Generation Genetic Studies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Ali Torkamani, Director, Genomics, Scripps Translational Science Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-6835
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Receive genetic risk information — Risk scores are provided by ResearchKit app.

SUMMARY:
Many conditions affecting health are caused by a combination of environment, behaviors, and genes. While individuals can alter some factors in their lives to reduce the chances of developing different diseases (e.g., not smoking cigarettes), the contribution from genetic risk encoded by DNA remains with people throughout their lives. Scientists are still trying to determine the entirety of genetic factors that influence disease, but for some conditions it has been shown that the factors identified thus far can begin to identify people at high to low genetic risk. Looking across the genome, scientists can calculate a cumulative genetic risk score - which can be used to rank genetic risk compared to other worldwide populations.

The goal of this study is to determine how genetic risk influences health decisions and other things that can be controlled in life. The first genetic risk score is calculated for coronary heart disease (CAD). CAD ultimately leads to heart attacks, heart failure and sometimes sudden cardiac death and is the main reason heart disease remains as the number one cause of death worldwide. Other researchers have shown that this genetic risk score can be used to identify people with low, intermediate, and high risk for coronary heart disease. It has also been shown that the use of statins (cholesterol lowering drugs) provides greater benefit and protection against heart attack for people with high genetic risk for coronary artery disease.

Leveraging the Apple ResearchKit and the ResearchKit linked 23andMe API, customers of 23andMe are able to provide researchers access to their genomic data. Participants will use the ResearchKit app to provide consent, view study information, answer surveys, and contact the study team.

Participants will be asked to complete 3 surveys. One before viewing genetic risk scores, one immediately after viewing scores, and one 6 months after viewing scores.

ELIGIBILITY:
Inclusion Criteria:

* Customer of 23andMe willing to share their 23andMe data
* User of Apple mobile device

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Initiation of Statin Therapy | 6 months
  Participant begins taking Statin as indicated by survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.